CLINICAL TRIAL: NCT06941259
Title: Effects of Combined Rectus Sheath and Ilioinguinal Nerve Block on Opioid Consumption in Hand-Assisted Laparoscopic Donor Nephrectomy Patients: A Randomized Controlled Double-Blind Prospective Study
Brief Title: Effects of Combined Rectus Sheath and Ilioinguinal Nerve Block on Opioid Consumption in HALDN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024.394.IRB1.046
Record Dates: First submitted 2025-01-30; First posted 2025-04-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-01

CONDITIONS: Regional Anesthesia Morbidity
Keywords: rectus sheath block; ilioinguinal nerve block; hand assisted donor nephrectomy
MeSH Terms: interventions — salicylhydroxamic acid; Anesthesia, Local; Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Group A: After patients anesthetized under general anaesthesia, a combined rectus sheath block and ilioinguinal nerve block will be applied with physiological saline.
  Group B: After patients anesthetized under general anaesthesia, a combined rectus sheath block and ilioinguinal nerve block will be applied with 0.25% bupivacaine.
Who Masked: Participant, Care Provider
Masking Description: The patient will be blind whether they receive local anaesthesia or physiological saline as the nerve block ingredient.
  The care providers will be blind to the solution when they are performing the regional anaesthesia.
  The care providers will be blind when they are monitoring the patient after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Sham (Sham Comparator): After the induction of general anaesthesia, the rectus sheath block and ilioinguinal nerve block will be performed to patients with a solution containing only physiological saline.
  Interventions: Procedure: Rectus sheath and ilioinguinal nerve block with physiological saline
- Group Block (Active Comparator): After the induction of general anaesthesia, the rectus sheath block and ilioinguinal nerve block will be performed to patients with a solution containing 0.25% bupivacaine.
  Interventions: Procedure: Rectus sheath and ilioinguinal nerve block with local anaesthesia

INTERVENTIONS:
Procedure: Rectus sheath and ilioinguinal nerve block with physiological saline — Rectus sheath and ilioinguinal nerve block without local anaesthesia
  Other Names: Group A (Sham)
  Arms: Group Sham
Procedure: Rectus sheath and ilioinguinal nerve block with local anaesthesia — Rectus sheath and ilioinguinal nerve block with local anaesthesia
  Other Names: Group B (Block)
  Arms: Group Block

SUMMARY:
The goal of this double-blind randomized control clinical trial is to investigate the effectiveness of regional anaesthesia blocks (rectus sheath block and ilioinguinal nerve block) on pain management in patients undergoing hand assisted laparoscopic donor nephrectomy surgery. The main question it aims to answer is:

Does combined rectus sheath block and ilioinguinal nerve block lower the amount of postoperative opioid consumption? Does reduced postoperative opioid consumption reduce the incidence of potential opioid related side effects? Does the application of nerve block affect length of hospital stay?

Researchers will compare patients who had nerve blocks with regional anaesthesia to a placebo group to see if total postoperative opioid consumption.

Participants will be randomly divided in two. Regional anaesthesia with local anaesthesia or a placebo will be performed. Patients will be followed 24 hours postoperatively to measure total opioid consumption.

Possible side effects, complications and length of hospital stay will be noted.

DETAILED DESCRIPTION:
In this study, it was planned to provide pain management after HALDN by applying a combined rectus sheath block and ilioinguinal nerve block. It is aimed to demonstrate the postoperative analgesic effectiveness of combined rectus sheath and ilioinguinal nerve block applied in addition to general anaesthesia in HALDN surgery. It was aimed to examine the amount of narcotic analgesic consumption in patients who received local anaesthetic for the first 24 hours after surgery. Regional anaesthesia applications with physiological saline, defined as 'Sham Block' in the literature, were preferred as the comparison group.

This method is a widely used comparison method and is used to obtain a double-blind study design.

ELIGIBILITY:
Inclusion Criteria:

* The donors reviewed by the transplant committee and deemed suitable for nephrectomy.
* Laparoscopic hand assisted donor nephrectomy operation is planned.

Exclusion Criteria:

* Allergy to any of the drugs to be used in treatment
* Patients using chronic narcotics or narcotic receptor agonists
* Patients with psychiatric disorders
* Patients with chronic organ failure
* Patients without end organ damage
* The patients who did not give consent
* Foreign national patients
* Patients with American Society of Anaesthesiologists (ASA) physical status classification score III and above

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-03-30 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 24 hours post-surgery
  Determination of the total amount of narcotic painkillers used during this period.

SECONDARY OUTCOMES:
Secondary Outcome | 24 hours post-surgery
  Numeric rating scale scores for pain after surgery. Numeric rating scale scores for pain of 1 being minimum amount of pain and 10 being the worse pain.
Secondary Outcome | 24 hours post-surgery
  Incidence of narcotic-related side effects
Secondary Outcome | through patient discharge postoperative, an average of 5 days postoperatively
  Length of hospital stay
Secondary Outcome | 1,3,6,12 hours post-surgery
  Determination of the total amount of narcotic painkillers used.
Secondary Outcome | 1,3,6,12 hours post-surgery
  Numeric rating scale scores for pain after surgery. Numeric rating scale scores for pain of 1 being minimum amount of pain and 10 being the worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Sincer, MD, Principal Investigator — Koç University
Locations (1):
- Koç University Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ozkalayci O, Karakaya MA, Yenigun Y, Cetin S, Darcin K, Akyollu B, Arpali E, Kocak B, Gurkan Y. Effects of erector spinae plane block on opioid consumption in patients undergoing hand-assisted laparoscopic donor nephrectomy: a randomized controlled trial. Minerva Anestesiol. 2024 Mar;90(3):154-161. doi: 10.23736/S0375-9393.23.17706-6. Epub 2024 Feb 2. PMID 38305014
- [Result] Gunaydin B, Ucar T, Arpali E, Akyollu B, Akinci S, Karatas C, Oztorun K, Kocak B. Hand-assisted laparoscopic donor nephrectomy: 1864 cases in 15 years of experience. Turk J Med Sci. 2022 Aug;52(4):1322-1328. doi: 10.55730/1300-0144.5438. Epub 2022 Aug 10. PMID 36326419

DOCUMENTS (1):
  • Informed Consent Form (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT06941259/ICF_000.pdf